CLINICAL TRIAL: NCT06281132
Title: A Randomized, Open-label, Single Dose, 4-period Replicate Crossover Study to Evaluate the Pharmacokinetic Profiles and Safety of CKD-341 in Healthy Volunteers Under Fasting Conditions
Brief Title: Clinical Trial to Compare and Evaluate the Safety and Pharmacokinetic After Oral Administration of CKD-341 and D956 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Chong Kun Dang Pharmaceutical (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: A126_03BE2316
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2024-05-28 (Actual); Status verified 2024-05

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — Tablets

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sequence 1 (Experimental): * Period 1: D956
  * Period 2: CKD-341
  * Period 3: D956
  * Period 4: CKD-341
  Interventions: Drug: CKD-341, D956
- Sequence 2 (Experimental): * Period 1: CKD-341
  * Period 2: D956
  * Period 3: CKD-341
  * Period 4: D956
  Interventions: Drug: CKD-341, D956

INTERVENTIONS:
Drug: CKD-341, D956 — A single dose of 1 tablet under fasting condition
  Other Names: PO, Tablet

SUMMARY:
The objective was to evaluate and compare the pharmacokinetic profiles and safety after administration of test drug (CKD-341) and reference drugs (D956) in healthy adults.

DETAILED DESCRIPTION:
A randomized, open-label, single dose, 4-period replicate crossover study in healthy adults under fasting conditions

ELIGIBILITY:
Inclusion Criteria:

1. Healthy adults aged between 19 to 55 years at the time of screening.
2. Individuals who had 18.0 kg/m2 ≤ Body Mass Index (BMI) < 30.5 kg/m2 and whose body weight was ≥ 55 kg.

   ☞ BMI = weight(kg) / height(m)2
3. Individuals without congenital/chronic diseases and without abnormal symptoms or diagnosis based on a medical examination within the last 3 years.
4. Individuals who were deemed to be appropriate as study subjects according to the laboratory tests (hematology, blood chemistry, urinalysis, serology, etc.), vital signs, 12-lead electrocardiogram (ECG), etc., performed at screening.
5. Individuals who signed an informed consent form approved by the Institutional Review Board (IRB) of Jeonbuk National University Hospital and who decided to participate voluntarily in the study after being fully informed of the study objective, contents, etc. prior to participation.
6. Individuals who consented to the use of reliable contraception (contraceptive methods other than hormones: use of condoms, intrauterine devices (IUD, IUS), tubal ligation, cervical cap, contraceptive diaphragm, etc.) during the clinical trial and not to donate sperm until 1 month after the last administration of investigational product(s).
7. Individuals with the ability and willingness to participate the entire study period.

Exclusion Criteria:

1. Individuals with medical evidence or a history (excluding a simple dental history of dental calculus, impacted tooth, wisdom tooth, etc.) of clinically significant hematological, renal, endocrine, respiratory, gastrointestinal(Active gastric ulcer), duodenal ulcer, etc.), urinary, cardiovascular (severe aortic valve stenosis, aArterial valve, mitral valve stenosis, obstructive hypertrophic cardiomyopathy, etc.), hepatic (severe hepatic impairment, etc.), psychiatric, neurologic, or immune diseases.
2. Individuals with a medical history of gastrointestinal diseases (e.g., esophageal disorders such as esophageal achalasia or esophagostenosis, Crohn's disease) or operations (excluding simple appendectomy, herniotomy, or tooth extraction) that may affect drug absorption.
3. Individuals with the following laboratory test result at screening:

   * ALT or AST > 2x the upper limit of the normal range
   * CK > 3x the upper limit of the normal range
   * eGFR <60 mL/min/1.73 m2 using CKD-EPI formula
4. Individuals with a history of regular alcohol consumption exceeding 210 g/week within 6 months prior to screening (1 drink (250 mL) of beer (5%) = 10 g; 1 drink (50 mL) of hard liquor (20%) = 8 g; 1 drink (125 mL) of wine (12%) = 12 g).
5. Individuals who smoked more than 20 cigarettes per day within 6 months prior to screening.
6. Individuals who had taken investigational product(s) from other clinical trials or bioequivalence studies within 6 months prior to the first administration of the investigational product(s).
7. Individuals with the following vital signs upon screening

   ☞ Systolic blood pressure ≥140 mmHg or <90 mmHg and/or a diastolic blood pressure ≥90 mmHg or <60 mmHg in sitting position.
8. Individuals with a medical history of significant alcohol or drug abuse within 1 year prior to the screening.
9. Individuals who had taken any drug(s) known as a strong inducer(s) or inhibitor(s) of drug-metabolizing enzymes within 30 days prior to the first administration of the investigational product(s).
10. Individuals who had taken prescription or nonprescription drugs within 10 days prior to the first administration of the investigational product(s).
11. Individuals who donated whole blood within 2 months or blood components within 1 month or have given blood transfusion within 1 month prior to the first administration of the investigational product(s).
12. Individuals with severe acute/chronic medical or psychological conditions, whose participation in the clinical trial and administration of the investigational products could increase the risk to the subjects or interfere with the interpretation of trial results.
13. Individuals with hypersensitivity to the investigational product(s), components of the investigational product(s), or dihydropyridine drugs, thiazide diuretics, or sulfonamide drugs, or hereditary issues of intolerance etc.
14. Patients with hereditary angioedema or with a history of angioedema when treated with ACE inhibitors or angiotensin II receptor antagonists.
15. Patients with shock.
16. Patients with anuria.
17. Patients with biliary obstructive disease.
18. Patients with diabetes or moderate to severe renal impairment who use aliskiren-containing preparations in combination.
19. Patients with severe heart failure.
20. Patients with Hypokalemia.
21. Patients with hyponatremia, hypercalcemia.
22. Patients with Hyperuricemia (with gout or uric acid stone).
23. Patients with Addison's syndrome.
24. Patients receiving lithium therapy.
25. Patients taking terfenadine or astemizole (can cause QT prolongation and ventricular arrhythmias).
26. Women who are pregnant or lactating.
27. Individuals who were deemed inappropriate to participate in the study by the investigator.

Ages: 19 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 51 (Actual)
Dates: Start 2024-03-22 (Actual); Primary Completion 2024-05-07 (Actual); Study Completion 2024-05-14 (Actual)

PRIMARY OUTCOMES:
area under curve(AUC) of CKD-341, D956 | Pre-dose(0 hour), post-dose 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hours
  Area under the CKD-341, D958 concentration in blood-time curve from zero to
Cmax of CKD-341, D956 | Pre-dose(0 hour), post-dose 0.25, 0.5, 0.75, 1, 1.25, 1.5, 1.75, 2, 3, 4, 5, 6, 8, 10, 12, 24, 48, 72 hours
  The maximum CKD-341, D956 concentration in blood sampling time

CONTACTS AND LOCATIONS:
Locations (1):
- Jeonbuk National University Hospital, Jeonju, South Korea

IPD SHARING:
Plan to Share IPD: No